CLINICAL TRIAL: NCT03394924
Title: A Phase 2 Dose Ranging, Randomized, Double Blind, Placebo-Controlled Study Evaluating the Safety, Tolerability, Pharmacokinetics and Efficacy of EDP-305 in Subjects With Primary Biliary Cholangitis (PBC) With or Without an Inadequate Response to Ursodeoxycholic Acid (UDCA)
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of EDP-305 in Subjects With Primary Biliary Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Collaborators: Pharmaceutical Research Associates (Other); Triangle Biostatistics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP 305-201
Record Dates: First submitted 2017-12-23; First posted 2018-01-09 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2020-06

CONDITIONS: Primary Biliary Cholangitis
Keywords: PBC; Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — EDP-305

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EDP-305 1 mg (Experimental): Subjects will take 2 tablets once a day orally for 12 weeks
  Interventions: Drug: EDP-305 1 mg
- EDP-305 2.5 mg (Experimental): Subjects will take 2 tablets once a day orally for 12 weeks
  Interventions: Drug: EDP-305 2.5 mg
- Placebo (Placebo Comparator): Subjects will take two tablets once a day orally for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-305 1 mg — Two tablets daily for 12 weeks
  Arms: EDP-305 1 mg
Drug: EDP-305 2.5 mg — Two tablets daily for 12 weeks
  Arms: EDP-305 2.5 mg
Drug: Placebo — Two tablets daily for 12 weeks
  Arms: Placebo

SUMMARY:
A randomized, double-blind study to assess the safety, tolerability, PK and efficacy of EDP-305 in subjects with primary biliary cholangitis

ELIGIBILITY:
Inclusion Criteria:

* An informed consent document signed and dated by the subject.
* Male and female subjects of any ethnic origin between the ages of 18 and 75 years, inclusive
* Male or female with a diagnosis of PBC by at least two of the following criteria:

  * History of ALP above ULN for at least six months
  * Positive Anti-Mitochondrial Antibodies (AMA) titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies)
* For subjects with no documented liver biopsy performed within 2 years, subjects must undergo a transient elastography (Fibroscan) showing liver stiffness < 14.0 kPA
* Must be on a stable dose of UDCA12-20 mg/kg/day for at least 6 months prior to Screening or intolerant of UDCA in the opinion of the Investigator (no UDCA for at least 12 weeks prior to Screening)
* Alkaline Phosphatase (ALP) ≥ 1.67 × ULN and/or total bilirubin >ULN but < 2×ULN (<2.4 mg/dL)
* Subjects must have Screening laboratory values for Hepatitis B surface antigen (HBsAg), anti-HCV antibodies and HCV RNA negative and Human Immunodeficiency Virus (HIV) 1 and 2 antibodies (Ab) as seronegative. Note: subjects previously infected by chronic hepatitis C and treated with direct acting antivirals (DAAs) with sustained virologic response (SVR) for at least 3 years will be allowed.
* Female subjects of childbearing potential must agree to use two effective methods of contraception from the date of Screening until 90 days after the last dose of EDP-305.
* All male participants who have not had a vasectomy must use effective contraception from Day -1 to 90 days after their last dose of study drug.
* Male subjects must agree to refrain from sperm donation from the date of Screening until 90 days after their last dose of study drug
* Screening body mass index (BMI) of ≥18 kg/m2
* Subject must be willing and able to adhere to the assessments, visit schedule, prohibitions and restrictions, as described in this protocol

Exclusion Criteria:

* Laboratory Screening Results:

  * AST >5 x ULN
  * ALT >5 x ULN
  * Patients with Gilbert's syndrome will not be allowed due to interpretability of bilirubin levels
  * Total white blood cells (WBC) <3000 cells/mm3
  * Absolute neutrophil count (ANC) <1500 cells/mm3
  * Platelet count <140,000/mm3
  * Prothrombin time (international normalized ratio, INR) >1.2
  * Serum creatinine >2 mg/dL or creatinine clearance <60 mL/min (based on Cockroft-Gault Method)
* Suspected to have relevant nonalcoholic fatty liver disease (NAFLD) as based on the judgment of the Investigator at Screening
* Use of immunosuppressants known to have an effect on the liver of patients with PBC (eg, colchicine, methotrexate, azathioprine, or systemic steroids) in the three months preceding screening
* Current use of fibrates, including fenofibrates. Note: Subjects who discontinued fibrates for at least 3 months before Screening can participate
* Use of an experimental treatment for PBC within the past 6 months
* Co-existing liver or biliary diseases, such as primary sclerosing cholangitis, choledocholithiasis, acute or chronic hepatitis, autoimmune hepatitis, alcoholic liver disease, nonalcoholic steatohepatitis (NASH), acute infection of bile duct system or gall bladder, history of gastrointestinal bleeding (secondary to portal hypertension), cirrhosis, cholangiocarcinoma diagnosed or suspected liver cancers
* Cirrhosis with or without complications, including history or presence of: spontaneous bacterial peritonitis, hepatocellular carcinoma
* Hepatorenal syndrome (type I or II) or Screening serum creatinine > 2 mg/dL (178 μmol/L)
* Prior variceal hemorrhage, uncontrolled encephalopathy, Child-Pugh Class A, B and C, esophageal varices, or refractory ascites within the previous 6 months of Screening (defined as date informed consent signed)
* Medical conditions that may cause nonhepatic increases in ALP (e.g., Paget's disease)
* Use of a new statin regimen from Screening and throughout study duration. NOTE: Subjects on a stable dose of statins for at least 3 months prior to Screening are allowed. No dose modification during the study will be allowed.
* Use of immunosuppressants (eg, systemic corticosteroids) for more than 2 consecutive weeks in duration within 1 year prior to Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (86):
- United States (40):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Arkansas Diagnostic Center, Little Rock, Arkansas
  - Texas Clinical Research Institute, Little Rock, Arkansas
  - Southern California Research Center, Coronado, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Liver Research Institue, Pasadena, California
  - Pasadena Liver Center, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - California Pacific Medical Center, San Francisco, California
  - South Denver Gastroenterology - Swedish Medical Center Office, Englewood, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - University of Miami Leonard M. Miller School of Medicine, Miami, Florida
  - Consultative Gastroenterology, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Louisiana Research Center, Shreveport, Louisiana
  - Mercy Medical Center-McAuley Plaza, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Digestive Disease Associates, Catonsville, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - CHI Health, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Northwell Health, Manhasset, New York
  - Concorde Medical Group, New York, New York
  - Mount Sinai Beth Isreal, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center - Bronx, The Bronx, New York
  - University of Pittsburgh Medical Center - Center for Liver Disease, Pittsburgh, Pennsylvania
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Liver Consultants of Texas, Dallas, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - Liver Institute of Virginia-Bremo, Richmond, Virginia
  - Swedish First Hill Campus, Seattle, Washington
  - University of Washington, Seattle, Washington
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Linear Clinical Research, Perth, Western Australia
- Austria (3):
  - Klinikum Klagenfurt Am Wörthersee, Klagenfurt, Carinthia
  - Medizinische Universität Innsbruck, Innsbruck, Tyrol
  - Klinikum Wels-Grieskirchen, Wels, Upper Austria
- Belgium (3):
  - CHU de Liège, Cardiology Dept., Liège, Liege
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Universitair Ziekenhuis Gent, Ghent, Oost-vlaanderen
- Canada (3):
  - London Health Sciences Centre University Hospital, London, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Liver Center, Toronto, Ontario
- France (8):
  - Nouvel Hôpital Civil, Strasbourg, Alsace
  - Hôpital Haut-Lévêque, Pessac, Aquitaine
  - Hôpital de la Croix Rousse, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire de Lille, Lille, Hauts-de-France
  - Hôpital Saint-Eloi, Montpellier, Languedoc-roussillon
  - Centre Hospitalier Universitaire Amines-Picardie Hôpital Sud, Amiens, Picardie
  - Hôpital Saint-Antoine, Paris, Île-de-France Region
  - Hôpital Paul Brousse, Villejuif, Île-de-France Region
- Germany (7):
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Charité Universitätsmedizin Berlin, Berlin
- Netherlands (3):
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Leiden Universitair Medisch Centrum, Leiden, South Holland
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (8):
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Universidad de Valladolid - Hospital Universitario Rio Hortega, Valladolid
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - The Leeds Teaching Hospitals NHS Trust, Leeds, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, England
  - Queen's Medical Centre - Nottingham, Nottingham, England
  - Portsmouth Hospitals NHS Trust, Portsmouth, England
  - NHS Lothian, Edinburgh, Scotland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial included 68 participants from 43 sites in Australia, Canada, Europe and the United States from December 2017 to January 2020.
Pre-assignment Details: 132 participants were screened, 64 of which were screen failures. The remaining 68 were enrolled and received trial treatment.
Groups:
- EDP-305 1 mg: Participants took EDP-305 1 milligrams (mg) as an oral tablet once daily for 12 weeks.
- EDP-305 2.5 mg: Participants took EDP-305 2.5 mg as an oral tablet once daily for 12 weeks.
- Placebo: Participants received an oral placebo matching EDP-305 once daily for 12 weeks.
Period: Overall Study
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Started | 31 | 28 | 9
Completed | 28 | 22 | 9
Not Completed | 3 | 6 | 0
Not completed — Adverse Event | 0 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Did not meet all inclusion criteria | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- EDP-305 1 mg: Participants took EDP-305 1 mg as an oral tablet once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo | Total
Number analyzed (Participants) | 31 | 28 | 9 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (8.61) | 54.9 (10.92) | 56.9 (8.49) | 56.3 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 27 | 9 | 67
  Male | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 5
  Not Hispanic or Latino | 27 | 25 | 9 | 61
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 27 | 9 | 64
  All other races | 3 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 16 | 12 | 2 | 30
  Canada | 1 | 1 | 1 | 3
  Australia | 2 | 1 | 2 | 5
  Spain | 3 | 2 | 2 | 7
  United Kingdom | 6 | 6 | 1 | 13
  Austria | 0 | 2 | 0 | 2
  Belgium | 0 | 1 | 0 | 1
  France | 0 | 1 | 0 | 1
  Germany | 2 | 1 | 1 | 4
  Netherlands | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least a 20% Reduction in Alkaline Phosphatase (ALP) or Normalization of ALP at Week 12 Compared to Baseline
Description: Percent change was calculated as [(ALP at Week 12 - ALP at Baseline)/ALP at Baseline] *100. The participant was considered to have successfully achieved a 20% reduction in ALP if the result was ≤-20. The participant was considered to have successfully achieved ALP normalization if ALP was abnormal at Baseline and normal at Week 12.
Time Frame: Baseline and Week 12
Population: Full Efficacy Population: All subjects who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
percentage of participants | 45.2 | 46.4 | 11.1
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Test type: Superiority; p = 0.106, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 5.6, 95% CI 2-sided [0.6 to 52]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Test type: Superiority; p = 0.063, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 7, 95% CI 2-sided [0.75 to 65.22]

2. Secondary Outcome: Percentage of Participants With a Treatment-Emergent Adverse Event (TEAE) During On-Treatment Period
Description: An adverse event (AE) was defined as any event, side effect, or untoward medical occurrence in a subject enrolled in a clinical trial whether or not it is considered to have a causal relationship to the study drug. A TEAE was an AE that first occurred or began previous to and worsened on or after the first dose date and before the last dose date +7 days.
Time Frame: Up to approximately Week 12
Population: Full Efficacy Population: All subjects who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Percentage of participants | 71.0 | 89.3 | 88.9

3. Secondary Outcome: Percentage of Participants With a Treatment-Emergent Serious Adverse Event (SAE) During On-Treatment Period
Description: A SAE is any untoward medical occurrence at any dose that results in death, is a life-threatening event, requires inpatient hospitalization or prolonged hospitalization of an existing hospitalization, results in permanent or prolonged disability or incapacity, is a congenital anomaly or birth defect in the offspring of a study subjects, or is a medically important event.
Time Frame: Up to approximately Week 12
Population: Full Efficacy Population: All subjects who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Percentage of participants | 3.2 | 7.1 | 0

4. Secondary Outcome: Percentage of Participants Who Stopped Study Treatment Due to a Treatment-Emergent Adverse Event (TEAE) During On-Treatment Period
Description: as for outcome 2
Time Frame: Up to approximately Week 12
Population: Full Efficacy Population: All subjects who received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Percentage of participants | 3.2 | 17.9 | 0

5. Secondary Outcome: Change From Baseline to Week 12 in Total, Conjugated and Unconjugated Bilirubin
Description: The data presented below was measured using least square mean change from baseline.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
μmol/L
  Total | -0.04 [-0.93 to 0.86] | -0.31 [-1.35 to 0.74] | -0.50 [-2.13 to 1.12]
  Conjugated | -0.55 [-1.03 to -0.06] | -0.51 [-1.08 to 0.06] | 0.13 [-0.75 to 1.00]
  Unconjugated | 0.71 [-0.02 to 1.44] | 0.22 [-0.61 to 1.06] | -0.50 [-1.81 to 0.81]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for total bilirubin; Test type: Superiority; p = 0.616, ANCOVA; Least squares mean difference = 0.47, 95% CI 2-sided [-1.39 to 2.32]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for total bilirubin; Test type: Superiority; p = 0.844, ANCOVA; Least squares mean difference = 0.19, 95% CI 2-sided [-1.78 to 2.16]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for conjugated bilirubin; Test type: Superiority; p = 0.18, ANCOVA; Least squares mean difference = -0.67, 95% CI 2-sided [-1.67 to 0.32]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for conjugated bilirubin; Test type: Superiority; p = 0.239, ANCOVA; Least squares mean difference = -0.64, 95% CI 2-sided [-1.71 to 0.44]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for unconjugated bilirubin; Test type: Superiority; p = 0.116, ANCOVA; Least squares mean difference = 1.21, 95% CI 2-sided [-0.31 to 2.73]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for unconjugated bilirubin; Test type: Superiority; p = 0.36, ANCOVA; Least squares mean difference = 0.72, 95% CI 2-sided [-0.84 to 2.28]

6. Secondary Outcome: Change From Baseline to Week 12 in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), and Gamma Glutamyl Transferase (GGT)
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: U/L
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
U/L
  ALT: number analyzed (Participants) | 28 | 21 | 9
  ALT | -17.35 [-24.45 to -10.25] | -13.14 [-21.58 to 4.71] | 8.20 [-4.61 to 21.02]
  AST: number analyzed (Participants) | 28 | 21 | 9
  AST | -12.08 [-17.49 to -6.68] | -11.51 [-17.91 to -5.10] | 9.33 [-0.43 to 19.09]
  GGT: number analyzed (Participants) | 28 | 21 | 9
  GGT | -95.91 [-114.12 to -77.70] | -124.55 [-146.00 to -103.11] | -9.42 [-42.19 to 23.35]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for ALT; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = -25.55, 95% CI 2-sided [-40.07 to -11.04]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for ALT; Test type: Superiority; p = 0.009, ANCOVA; Least squares mean difference = -21.35, 95% CI 2-sided [-37.1 to -5.6]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for AST; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = -21.42, 95% CI 2-sided [-32.48 to -10.35]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for AST; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = -20.84, 95% CI 2-sided [-32.8 to -8.87]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for GGT; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = -86.49, 95% CI 2-sided [-123.78 to -49.21]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for GGT; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = -115.13, 95% CI 2-sided [-155.04 to -75.22]

7. Secondary Outcome: Change From Baseline to Week 12 in Noninvasive Liver Fibrosis Markers: Enhanced Liver Fibrosis (ELF) Panel and N-terminal Type III Collagen Propeptide (PRO C3)
Description: The ELF panel included hyaluronic acid (HA), procollagen III amino terminal peptide (PIIINP), and tissue inhibitor of metalloproteinase 1 (TIMP 1). This endpoint also presents PRO C3 results.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/L
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
μg/L
  HA: number analyzed (Participants) | 28 | 21 | 9
  HA | 1.17 [-16.69 to 19.03] | -1.16 [-22.20 to 19.87] | 27.83 [-4.20 to 59.86]
  PIIINP: number analyzed (Participants) | 28 | 21 | 9
  PIIINP | -0.08 [-1.28 to 1.11] | -0.77 [-2.20 to 0.65] | 3.01 [0.72 to 5.30]
  TIMP 1: number analyzed (Participants) | 28 | 21 | 9
  TIMP 1 | -16.29 [-32.31 to -0.27] | -20.90 [-39.58 to -2.22] | 25.66 [-3.64 to 54.97]
  PRO C3: number analyzed (Participants) | 19 | 18 | 8
  PRO C3 | -0.67 [-4.97 to 3.63] | 2.33 [-2.31 to 6.96] | 9.06 [2.16 to 15.95]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for HA; Test type: Superiority; p = 0.148, ANCOVA; Least squares mean difference = -26.66, 95% CI 2-sided [-63.1 to 9.79]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for HA; Test type: Superiority; p = 0.142, ANCOVA; Least squares mean difference = -28.99, 95% CI 2-sided [-68.02 to 10.05]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for PIIINP; Test type: Superiority; p = 0.02, ANCOVA; Least squares mean difference = -3.09, 95% CI 2-sided [-5.68 to -0.51]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for PIIINP; Test type: Superiority; p = 0.009, ANCOVA; Least squares mean difference = -3.79, 95% CI 2-sided [-6.6 to -0.97]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for TIMP 1; Test type: Superiority; p = 0.015, ANCOVA; Least squares mean difference = -41.96, 95% CI 2-sided [-75.47 to -8.44]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for TIMP 1; Test type: Superiority; p = 0.011, ANCOVA; Least squares mean difference = -46.56, 95% CI 2-sided [-81.91 to -11.21]
Statistical Analysis 7: Comparison: EDP-305 1 mg vs Placebo; Analysis for PRO C3; Test type: Superiority; p = 0.018, ANCOVA; Least squares mean difference = -9.73, 95% CI 2-sided [-17.7 to -1.75]
Statistical Analysis 8: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for PRO C3; Test type: Superiority; p = 0.125, ANCOVA; Least squares mean difference = -6.73, 95% CI 2-sided [-15.41 to 1.95]

8. Secondary Outcome: Change From Baseline to Week 12 in Noninvasive Liver Fibrosis Markers: AST to Platelet Ratio Index (APRI) Score
Description: APRI was calculated as ([AST level/AST upper limit of normal]/[Platelet count 1^09/L])×100. AST is aspartate aminotransferase. The aspartate transaminase to platelet ratio index (APRI) is used to assess liver fibrosis in participants with chronic liver disease. Scores range from 0 to ≥ 2.0, with scores < 0.5 predictive of no liver fibrosis; scores >1.5 significant fibrosis; and scores > 2.0 indicative of cirrhosis. A negative change from baseline indicates a decrease in fibrosis.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Index
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 24 | 20 | 8
Index | -0.16 [-0.25 to 0.06] | -0.12 [-0.23 to 0.01] | 0.22 [0.05 to 0.38]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = -0.37, 95% CI 2-sided [-0.56 to -0.18]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Test type: Superiority; p = 0.002, ANCOVA; Least squares mean difference = -0.33, 95% CI 2-sided [-0.54 to -0.13]

9. Secondary Outcome: Change From Baseline to Week 12 in Noninvasive Liver Fibrosis Markers: Fibrosis-4 (FIB-4) Score
Description: Fibrosis-4 is the ratio of age in years and aminotransferase to platelet count. It is a non-invasive hepatic fibrosis index score that is calculated using formula: FIB-4 = (Age [years] x AST [U/L]) / (platelets [10^9/L] x (square root of ALT [U/L])). A FIB-4 index of < 1.45 indicates no or moderate fibrosis and an index of > 3.25 indicates extensive fibrosis/cirrhosis. A positive change from Baseline indicates increased fibrosis.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Index
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 24 | 20 | 8
Index | -0.14 [-0.29 to 0.01] | -0.05 [-0.22 to 0.11] | 0.21 [-0.06 to 0.47]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Test type: Superiority; p = 0.026, ANCOVA; Least squares mean difference = -0.35, 95% CI 2-sided [-0.65 to -0.04]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Test type: Superiority; p = 0.104, ANCOVA; Least squares mean difference = -0.26, 95% CI 2-sided [-0.57 to 0.05]

10. Secondary Outcome: Change From Baseline to Week 12 in Fibrinogen and C Reactive Protein (CRP) Levels
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
mg/dL
  Fibrinogen: number analyzed (Participants) | 28 | 20 | 9
  Fibrinogen | 16.28 [-5.39 to 37.95] | 41.25 [15.56 to 66.93] | 9.47 [-28.82 to 47.76]
  CRP: number analyzed (Participants) | 27 | 21 | 8
  CRP | -0.57 [-1.62 to 0.49] | -2.69 [-3.89 to -1.50] | 0.41 [-1.53 to 2.34]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for fibrinogen; Test type: Superiority; p = 0.757, ANCOVA; Least squares mean difference = 6.81, 95% CI 2-sided [-37.17 to 50.78]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for fibrinogen; Test type: Superiority; p = 0.174, ANCOVA; Least squares mean difference = 31.77, 95% CI 2-sided [-14.42 to 77.97]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for CRP; Test type: Superiority; p = 0.378, ANCOVA; Least squares mean difference = -0.98, 95% CI 2-sided [-3.18 to 1.23]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for CRP; Test type: Superiority; p = 0.008, ANCOVA; Least squares mean difference = -3.1, 95% CI 2-sided [-5.38 to -0.83]

11. Secondary Outcome: Change From Baseline to Week 12 in Interleukin (IL) and Tumor Necrosis Factor (TNF) Levels
Description: For IL, both IL6 and IL1β variants were analysed. For TNF, both TNF α and TNF β (also known as lymphotoxin alpha) variants were analyzed.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/L
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
ng/L
  IL6: number analyzed (Participants) | 27 | 21 | 9
  IL6 | 0.73 [-0.97 to 2.43] | -2.10 [-4.03 to -0.17] | 0.39 [-2.57 to 3.34]
  IL1β: number analyzed (Participants) | 28 | 21 | 9
  IL1β | NA [NA to NA] — LS mean not computable as all analysed results were below limit of detection. | NA [NA to NA] — LS mean not computable as all analysed results were below limit of detection. | NA [NA to NA] — LS mean not computable as all analysed results were below limit of detection.
  TNF α: number analyzed (Participants) | 28 | 21 | 9
  TNF α | -0.15 [-0.38 to 0.09] | -0.01 [-0.28 to 0.25] | 0.39 [-0.03 to 0.81]
  TNF β: number analyzed (Participants) | 19 | 18 | 8
  TNF β | NA [NA to NA] — LS mean not computable as all analysed results were below limit of detection. | NA [NA to NA] — LS mean not computable as all analysed results were below limit of detection. | NA [NA to NA] — LS mean not computable as all analysed results were below limit of detection.
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for IL6; Test type: Superiority; p = 0.841, ANCOVA; Least squares mean difference = 0.34, 95% CI 2-sided [-3.07 to 3.76]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for IL6; Test type: Superiority; p = 0.163, ANCOVA; Least squares mean difference = -2.49, 95% CI 2-sided [-6.01 to 1.04]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for TNF α; Test type: Superiority; p = 0.03, ANCOVA; Least squares mean difference = -0.53, 95% CI 2-sided [-1.02 to -0.05]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for TNF α; Test type: Superiority; p = 0.11, ANCOVA; Least squares mean difference = -0.4, 95% CI 2-sided [-0.9 to 0.09]

12. Secondary Outcome: Change From Baseline to Week 12 in Haptoglobin and Alpha2 Macroglobulin Levels
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/L
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
g/L
  Haptoglobin: number analyzed (Participants) | 28 | 21 | 9
  Haptoglobin | -0.14 [-0.27 to -0.01] | -0.18 [-0.33 to -0.03] | -0.15 [-0.38 to 0.08]
  Alpha2 Macroglobulin: number analyzed (Participants) | 28 | 21 | 9
  Alpha2 Macroglobulin | -0.02 [-0.09 to 0.05] | -0.00 [-0.08 to 0.08] | 0.02 [-0.11 to 0.15]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for haptoglobin; Test type: Superiority; p = 0.944, ANCOVA; Least squares mean difference = 0.01, 95% CI 2-sided [-0.25 to 0.27]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for haptoglobin; Test type: Superiority; p = 0.83, ANCOVA; Least squares mean difference = -0.03, 95% CI 2-sided [-0.3 to 0.24]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for alpha2 macroglobulin; Test type: Superiority; p = 0.546, ANCOVA; Least squares mean difference = -0.04, 95% CI 2-sided [-0.19 to 0.1]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for alpha2 macroglobulin; Test type: Superiority; p = 0.785, ANCOVA; Least squares mean difference = -0.02, 95% CI 2-sided [-0.18 to 0.13]

13. Secondary Outcome: Change From Baseline to Week 12 in Triglycerides (TG), Total Cholesterol (TC), High Density Lipoprotein Cholesterol (HDL-C), Low Density Lipoprotein Cholesterol (LDL-C)
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
mmol/L
  TG: number analyzed (Participants) | 28 | 21 | 9
  TG | -0.13 [-0.25 to -0.00] | 0.01 [-0.13 to 0.16] | 0.05 [-0.17 to 0.27]
  TC: number analyzed (Participants) | 28 | 21 | 9
  TC | -0.47 [-0.80 to -0.14] | -0.46 [-0.85 to -0.08] | 0.17 [-0.42 to 0.76]
  HDL-C: number analyzed (Participants) | 28 | 21 | 9
  HDL-C | -0.16 [-0.31 to -0.02] | -0.46 [-0.62 to -0.30] | -0.24 [-0.49 to 0.01]
  LDL-C: number analyzed (Participants) | 28 | 21 | 9
  LDL-C | -0.21 [-0.47 to 0.05] | -0.01 [-0.31 to 0.29] | 0.29 [-0.19 to 0.76]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for TG; Test type: Superiority; p = 0.176, ANCOVA; Least squares mean difference = -0.17, 95% CI 2-sided [-0.43 to 0.08]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for TG; Test type: Superiority; p = 0.783, ANCOVA; Least squares mean difference = -0.04, 95% CI 2-sided [-0.3 to 0.23]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for TC; Test type: Superiority; p = 0.061, ANCOVA; Least squares mean difference = -0.64, 95% CI 2-sided [-1.31 to 0.03]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for TC; Test type: Superiority; p = 0.08, ANCOVA; Least squares mean difference = -0.63, 95% CI 2-sided [-1.34 to 0.08]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for HDL-C; Test type: Superiority; p = 0.584, ANCOVA; Least squares mean difference = 0.08, 95% CI 2-sided [-0.21 to 0.37]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for HDL-C; Test type: Superiority; p = 0.148, ANCOVA; Least squares mean difference = -0.22, 95% CI 2-sided [-0.51 to 0.08]
Statistical Analysis 7: Comparison: EDP-305 1 mg vs Placebo; Analysis for LDL-C; Test type: Superiority; p = 0.074, ANCOVA; Least squares mean difference = -0.5, 95% CI 2-sided [-1.04 to 0.05]
Statistical Analysis 8: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for LDL-C; Test type: Superiority; p = 0.304, ANCOVA; Least squares mean difference = -0.3, 95% CI 2-sided [-0.87 to 0.28]

14. Secondary Outcome: Change From Baseline to Week 12 in Domain and Total Scores on the 5D-Itch Scale
Description: The 5D-Itch scale is a multidimensional questionnaire completed by participants to quantify the magnitude of pruritus, assessed considering the past 2 weeks. Scale range is 1 to 5 covering five dimensions: duration (1=Less than 6 hrs/day to 5=All day), degree (1=Not present to 5=Unbearable), direction (1=Completely resolved to 5=Getting worse), disability (for Sleep rated as 1=Never affects sleep to 5=Delays falling asleep and frequently wakes me up at night; for Leisure/Social, Housework/Errands and Work/School rated as 1=Never affects activity to 5=Always affects activity), and distribution (assess if itching is present in 16 body locations, scored as 1=present at 0-2 locations to 5=present at 14-16 locations). Total scores (including highest disability score obtained from any of the daily activities) ranged between 5 and 25 where higher scores indicated more severe itching. Negative change scores indicate improvement from the baseline score.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Scores on a scale
  Duration: number analyzed (Participants) | 24 | 21 | 8
  Duration | 0.01 [-0.27 to 0.29] | 0.41 [0.11 to 0.71] | -0.24 [-0.73 to 0.25]
  Degree: number analyzed (Participants) | 26 | 21 | 9
  Degree | 0.00 [-0.25 to 0.26] | 0.65 [0.37 to 0.93] | -0.53 [-0.96 to 0.10]
  Direction: number analyzed (Participants) | 25 | 21 | 9
  Direction | -0.63 [-1.12 to -0.15] | 0.36 [-0.17 to 0.90] | -0.65 [-1.46 to 0.16]
  Disability: number analyzed (Participants) | 26 | 21 | 9
  Disability | -0.24 [-0.63 to 0.15] | 0.85 [0.42 to 1.28] | -0.61 [-1.28 to 0.05]
  Distribution: number analyzed (Participants) | 26 | 21 | 9
  Distribution | 0.07 [-0.32 to 0.45] | 0.81 [0.38 to 1.24] | -0.42 [-1.08 to 0.24]
  Total: number analyzed (Participants) | 24 | 21 | 8
  Total | -0.95 [-2.29 to 0.39] | 3.19 [1.74 to 4.64] | -3.16 [-5.50 to -0.82]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for duration; Test type: Superiority; p = 0.378, ANCOVA; Least squares mean difference = 0.25, 95% CI 2-sided [-0.32 to 0.82]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for duration; Test type: Superiority; p = 0.03, ANCOVA; Least squares mean difference = 0.65, 95% CI 2-sided [0.07 to 1.23]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for degree; Test type: Superiority; p = 0.036, ANCOVA; Least squares mean difference = 0.53, 95% CI 2-sided [0.04 to 1.03]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for degree; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = 1.18, 95% CI 2-sided [0.67 to 1.69]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for direction; Test type: Superiority; p = 0.971, ANCOVA; Least squares mean difference = 0.02, 95% CI 2-sided [-0.92 to 0.96]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for direction; Test type: Superiority; p = 0.042, ANCOVA; Least squares mean difference = 1.01, 95% CI 2-sided [0.04 to 1.99]
Statistical Analysis 7: Comparison: EDP-305 1 mg vs Placebo; Analysis for disability; Test type: Superiority; p = 0.336, ANCOVA; Least squares mean difference = 0.37, 95% CI 2-sided [-0.4 to 1.14]
Statistical Analysis 8: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for disability; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = 1.46, 95% CI 2-sided [0.67 to 2.26]
Statistical Analysis 9: Comparison: EDP-305 1 mg vs Placebo; Analysis for distribution; Test type: Superiority; p = 0.214, ANCOVA; Least squares mean difference = 0.48, 95% CI 2-sided [-0.29 to 1.25]
Statistical Analysis 10: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for distribution; Test type: Superiority; p = 0.003, ANCOVA; Least squares mean difference = 1.23, 95% CI 2-sided [0.44 to 2.02]
Statistical Analysis 11: Comparison: EDP-305 1 mg vs Placebo; Analysis for total; Test type: Superiority; p = 0.103, ANCOVA; Least squares mean difference = 2.21, 95% CI 2-sided [-0.47 to 4.9]
Statistical Analysis 12: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for total; Test type: Superiority; p = 0.000, ANCOVA; Least squares mean difference = 6.35, 95% CI 2-sided [3.57 to 9.13]

15. Secondary Outcome: Change From Baseline to Week 12 in Visual Analog Score (VAS) for Itching
Description: An itch VAS (0-100mm) was used to record the intensity of the event. Participants drew a line on a scale corresponding to the maximum intensity of itch. Lines drawn towards the right of the line indicated greater itching and higher scores indicated more severe itching. Negative change from baseline indicates decrease in itching.
Time Frame: Baseline to Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 26 | 22 | 9
Scores on a scale | 0.55 [-8.35 to 9.44] | 13.64 [4.00 to 23.29] | -11.93 [-27.05 to 3.18]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Test type: Superiority; p = 0.16, ANCOVA; Least squares mean difference = 12.48, 95% CI 2-sided [-5.09 to 30.06]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Test type: Superiority; p = 0.006, ANCOVA; Least squares mean difference = 25.58, 95% CI 2-sided [7.67 to 43.48]

16. Secondary Outcome: Change From Baseline to Week 12 in Domain Scores on the Primary Biliary Cholangitis-40 (PBC-40) Quality of Life (QoL) Assessment
Description: The PBC-40 is a survey measuring health related quality of life in participants with PBC. The 40 questions from the PBC-40 questionnaire are scored from 1-5, with 5 representing the highest impact and 1 the lowest impact of PBC on the quality of life. Six domains were computed from the 40 questions: symptoms (score range 7-35), itch (0-15), fatigue (11-55), cognition (6-30), social (8-50) and emotional (1-15). Higher scores indicate worse quality of life and negative change scores indicate improvement from the baseline score.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Scores on a scale
  Symptoms: number analyzed (Participants) | 28 | 21 | 9
  Symptoms | -0.21 [-1.47 to 1.06] | -1.46 [-2.93 to 0.00] | -0.06 [-2.30 to 2.18]
  Itch: number analyzed (Participants) | 28 | 21 | 9
  Itch | 0.18 [-0.72 to 1.09] | 1.74 [0.69 to 2.78] | -1.73 [-3.33 to -0.13]
  Fatigue: number analyzed (Participants) | 28 | 21 | 9
  Fatigue | -0.36 [-2.58 to 1.86] | -0.22 [-2.79 to 2.34] | 0.10 [-3.82 to 4.01]
  Cognition: number analyzed (Participants) | 28 | 21 | 9
  Cognition | -0.21 [-1.46 to 1.04] | 0.82 [-0.63 to 2.27] | -0.48 [-2.66 to 1.71]
  Social: number analyzed (Participants) | 28 | 21 | 9
  Social | -0.38 [-2.22 to 1.46] | 0.96 [-1.17 to 3.08] | 1.73 [-1.52 to 4.99]
  Emotional: number analyzed (Participants) | 28 | 21 | 9
  Emotional | -0.77 [-1.54 to 0.01] | 0.23 [-0.68 to 1.13] | -0.15 [-1.52 to 1.22]
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for symptoms; Test type: Superiority; p = 0.908, ANCOVA; Least squares mean difference = -0.15, 95% CI 2-sided [-2.72 to 2.43]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for symptoms; Test type: Superiority; p = 0.298, ANCOVA; Least squares mean difference = -1.41, 95% CI 2-sided [-4.09 to 1.27]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for itch; Test type: Superiority; p = 0.042, ANCOVA; Least squares mean difference = 1.91, 95% CI 2-sided [0.07 to 3.76]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for itch; Test type: Superiority; p = 0.001, ANCOVA; Least squares mean difference = 3.47, 95% CI 2-sided [1.55 to 5.38]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for fatigue; Test type: Superiority; p = 0.839, ANCOVA; Least squares mean difference = -0.46, 95% CI 2-sided [-4.96 to 4.04]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for fatigue; Test type: Superiority; p = 0.891, ANCOVA; Least squares mean difference = -0.32, 95% CI 2-sided [-5.00 to 4.36]
Statistical Analysis 7: Comparison: EDP-305 1 mg vs Placebo; Analysis for cognition; Test type: Superiority; p = 0.834, ANCOVA; Least squares mean difference = 0.26, 95% CI 2-sided [-2.25 to 2.77]
Statistical Analysis 8: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for cognition; Test type: Superiority; p = 0.327, ANCOVA; Least squares mean difference = 1.3, 95% CI 2-sided [-1.33 to 3.92]
Statistical Analysis 9: Comparison: EDP-305 1 mg vs Placebo; Analysis for social; Test type: Superiority; p = 0.262, ANCOVA; Least squares mean difference = -2.12, 95% CI 2-sided [-5.86 to 1.62]
Statistical Analysis 10: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for social; Test type: Superiority; p = 0.69, ANCOVA; Least squares mean difference = -0.78, 95% CI 2-sided [-4.68 to 3.12]
Statistical Analysis 11: Comparison: EDP-305 1 mg vs Placebo; Analysis for emotional; Test type: Superiority; p = 0.433, ANCOVA; Least squares mean difference = -0.62, 95% CI 2-sided [-2.19 to 0.95]
Statistical Analysis 12: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for emotional; Test type: Superiority; p = 0.653, ANCOVA; Least squares mean difference = 0.37, 95% CI 2-sided [-1.28 to 2.03]

17. Secondary Outcome: Maximum Plasma Concentration (Cmax) of EDP-305 and Its Metabolites
Description: Metabolites of EDP-305 are EP-022571, EP-022572, and EP-022679.
Time Frame: Day 1 and Week 12: Pre-dose and 2, 6 and 8 hours post-dose
Population: Blood samples for Pharmacokinetic (PK) analysis were collected from a subset of study sites and included participants who received active study drug and had any measurable plasma concentration of study drug at any timepoint. Results are presented for participants that have data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- EDP-305 1 mg - Pharmacokinetic Substudy: Participants took EDP-305 1 mg as an oral tablet once daily for 12 weeks.
- EDP-305 2.5 mg - Pharmacokinetic Substudy: Participants took EDP-305 2.5 mg as an oral tablet once daily for 12 weeks.
Arm/Group | EDP-305 1 mg - Pharmacokinetic Substudy | EDP-305 2.5 mg - Pharmacokinetic Substudy
Number analyzed (Participants) | 5 | 6
ng/mL
  EDP-305 Day 1: number analyzed (Participants) | 5 | 5
  EDP-305 Day 1 | 15.4 (44.30) | 27.9 (54.19)
  EDP-305 Week 12: number analyzed (Participants) | 4 | 4
  EDP-305 Week 12 | 10.8 (67.77) | 50.4 (53.20)
  EP-022571 Day 1: number analyzed (Participants) | 5 | 5
  EP-022571 Day 1 | 0.5 (44.58) | 0.6 (61.81)
  EP-022571 Week 12: number analyzed (Participants) | 4 | 4
  EP-022571 Week 12 | 0.2 (59.57) | 1.3 (160.28)
  EP-022572 Day 1: number analyzed (Participants) | 5 | 5
  EP-022572 Day 1 | 0.5 (41.69) | 0.8 (38.27)
  EP-022572 Week 12: number analyzed (Participants) | 4 | 4
  EP-022572 Week 12 | 0.2 (41.74) | 1.6 (138.55)
  EP-022679 Day 1: number analyzed (Participants) | 5 | 5
  EP-022679 Day 1 | 0.8 (113.24) | 1.7 (115.17)
  EP-022679 Week 12: number analyzed (Participants) | 4 | 4
  EP-022679 Week 12 | 0.6 (147.81) | 10.9 (352.53)

18. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of EDP-305 and Its Metabolites
Description: Metabolites of EDP-305 are EP-022571, EP-022572, and EP-022679.
Time Frame: Day 1 and Week 12: Pre-dose and 2, 6 and 8 hours post-dose
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | EDP-305 1 mg - Pharmacokinetic Substudy | EDP-305 2.5 mg - Pharmacokinetic Substudy
Number analyzed (Participants) | 5 | 6
hours
  EDP-305 Day 1: number analyzed (Participants) | 5 | 5
  EDP-305 Day 1 | 6.00 [2.02 to 6.03] | 6.02 [2.00 to 8.00]
  EDP-305 Week 12: number analyzed (Participants) | 4 | 4
  EDP-305 Week 12 | 7.01 [6.00 to 8.02] | 6.01 [2.05 to 8.02]
  EP-022571 Day 1: number analyzed (Participants) | 5 | 5
  EP-022571 Day 1 | 2.00 [2.00 to 6.00] | 6.00 [2.00 to 6.10]
  EP-022571 Week 12: number analyzed (Participants) | 4 | 4
  EP-022571 Week 12 | 6.00 [2.00 to 6.00] | 4.00 [2.00 to 6.10]
  EP-022572 Day 1: number analyzed (Participants) | 5 | 5
  EP-022572 Day 1 | 2.00 [2.00 to 8.00] | 6.00 [2.00 to 6.10]
  EP-022572 Week 12: number analyzed (Participants) | 4 | 4
  EP-022572 Week 12 | 6.00 [6.00 to 8.00] | 4.00 [2.00 to 6.00]
  EP-022679 Day 1: number analyzed (Participants) | 5 | 5
  EP-022679 Day 1 | 6.00 [6.00 to 8.00] | 6.10 [2.00 to 8.00]
  EP-022679 Week 12: number analyzed (Participants) | 4 | 4
  EP-022679 Week 12 | 6.00 [6.00 to 8.00] | 6.00 [6.00 to 8.00]

19. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of EDP-305 and Its Metabolites
Description: Metabolites of EDP-305 are EP-022571, EP-022572, and EP-022679.
Time Frame: Day 1 and Week 12: Pre-dose and 2, 6 and 8 hours post-dose
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | EDP-305 1 mg - Pharmacokinetic Substudy | EDP-305 2.5 mg - Pharmacokinetic Substudy
Number analyzed (Participants) | 5 | 6
h*ng/mL
  EDP-305 Day 1: number analyzed (Participants) | 5 | 5
  EDP-305 Day 1 | 85.50 (51.57) | 95.30 (141.72)
  EDP-305 Week 12: number analyzed (Participants) | 4 | 4
  EDP-305 Week 12 | 67.60 (75.47) | 316.20 (42.34)
  EP-022571 Day 1: number analyzed (Participants) | 5 | 5
  EP-022571 Day 1 | 2.30 (37.32) | 2.00 (132.47)
  EP-022571 Week 12: number analyzed (Participants) | 4 | 4
  EP-022571 Week 12 | 0.90 (78.75) | 7.30 (154.62)
  EP-022572 Day 1: number analyzed (Participants) | 5 | 5
  EP-022572 Day 1 | 2.50 (32.37) | 2.90 (96.70)
  EP-022572 Week 12: number analyzed (Participants) | 4 | 4
  EP-022572 Week 12 | 1.20 (53.12) | 10.10 (148.55)
  EP-022679 Day 1: number analyzed (Participants) | 5 | 5
  EP-022679 Day 1 | 3.70 (109.30) | 5.00 (305.62)
  EP-022679 Week 12: number analyzed (Participants) | 4 | 4
  EP-022679 Week 12 | 3.00 (203.04) | 57.00 (343.47)

20. Secondary Outcome: Percentage Change From Baseline to Week 12 in Fibroblast Growth Factor 19 (FGF19), 7α-OH-4-cholesten-3-one (C4) and Bile Acid (BA) Concentrations
Description: FGF19 was measured in plasma. BA was measured in serum. C4 was measured in serum.
Time Frame: Baseline and Week 12
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Percentage change from baseline
  FGF19: number analyzed (Participants) | 26 | 20 | 7
  FGF19 | 28.10 (94.526) | 46.90 (76.667) | 39.83 (100.579)
  C4: number analyzed (Participants) | 26 | 20 | 7
  C4 | -18.066 (114.9959) | -61.960 (42.8603) | 39.839 (163.6265)
  BA: number analyzed (Participants) | 23 | 14 | 7
  BA | -21.79 (74.581) | -15.79 (112.934) | 3.17 (48.656)
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for FGF19; Test type: Superiority; p = 0.971, ANCOVA; Least squares mean difference = 1.34, 95% CI 2-sided [-71.51 to 74.18]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for FGF19; Test type: Superiority; p = 0.882, ANCOVA; Least squares mean difference = 5.54, 95% CI 2-sided [-68.86 to 79.95]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for C4; Test type: Superiority; p = 0.242, ANCOVA; Least squares mean difference = -51.66, 95% CI 2-sided [-139.27 to 35.96]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for C4; Test type: Superiority; p = 0.042, ANCOVA; Least squares mean difference = -94.3, 95% CI 2-sided [-184.85 to -3.75]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for BA; Test type: Superiority; p = 0.52, ANCOVA; Least squares mean difference = -24.57, 95% CI 2-sided [-101.03 to 51.89]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for BA; Test type: Superiority; p = 0.672, ANCOVA; Least squares mean difference = -17.96, 95% CI 2-sided [-103.07 to 67.16]

21. Secondary Outcome: Percentage Change From Baseline to Week 12 in AUC0-8 and AUC2-8 of Fibroblast Growth Factor 19 (FGF19), 7α-OH-4-cholesten-3-one (C4) and Bile Acid (BA)
Description: AUC0-8 is area under the biomarker concentration-time curve from time zero to 8 hours. AUC2-8 is area under the biomarker concentration-time curve from 2 hours to 8 hours. FGF19 was measured in plasma. BA was measured in serum. C4 was measured in serum.
Time Frame: Day 1 and Week 12: Pre-dose and 2, 6 and 8 hours post-dose
Population: Results are presented for participants from the Full Efficacy Population that have data available for analysis.
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
Number analyzed (Participants) | 31 | 28 | 9
Percentage change from baseline
  FGF19 AUC0-8: number analyzed (Participants) | 4 | 2 | 1
  FGF19 AUC0-8 | 24.9 (68.90) | 25.0 (71.72) | -25.9 (NA) — SD not computable as only 1 participant was analysed.
  FGF19 AUC 2-8: number analyzed (Participants) | 5 | 2 | 1
  FGF19 AUC 2-8 | 7.8 (86.25) | 18.9 (66.35) | -25.3 (NA) — SD not computable as only 1 participant was analysed.
  C4 AUC0-8: number analyzed (Participants) | 4 | 1 | 1
  C4 AUC0-8 | 3.7 (51.74) | 100.0 (NA) — SD not computable as only 1 participant was analysed. | 138.2 (NA) — SD not computable as only 1 participant was analysed.
  C4 AUC2-8: number analyzed (Participants) | 5 | 1 | 1
  C4 AUC2-8 | -9.2 (66.30) | -100.0 (NA) — SD not computable as only 1 participant was analysed. | 122.5 (NA) — SD not computable as only 1 participant was analysed.
  BA AUC0-8: number analyzed (Participants) | 4 | 2 | 4
  BA AUC0-8 | -20.7 (74.80) | -51.5 (41.06) | -26.1 (NA) — SD not computable as only 1 participant was analysed.
  BA AUC2-8: number analyzed (Participants) | 5 | 2 | 1
  BA AUC2-8 | -33.6 (76.26) | -42.8 (56.77) | -24.4 (NA) — SD not computable as only 1 participant was analysed.
Statistical Analysis 1: Comparison: EDP-305 1 mg vs Placebo; Analysis for FGF19 AUC0-8; Test type: Superiority; p = 0.611, ANCOVA; Least squares mean difference = 44.54, 95% CI 2-sided [-205.97 to 295.06]
Statistical Analysis 2: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for FGF19 AUC0-8; Test type: Superiority; p = 0.819, ANCOVA; Least squares mean difference = -29.98, 95% CI 2-sided [-411.28 to 351.31]
Statistical Analysis 3: Comparison: EDP-305 1 mg vs Placebo; Analysis for FGF19 AUC2-8; Test type: Superiority; p = 0.818, ANCOVA; Least squares mean difference = 24.41, 95% CI 2-sided [-251.92 to 300.74]
Statistical Analysis 4: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for FGF19 AUC2-8; Test type: Superiority; p = 0.948, ANCOVA; Least squares mean difference = -10.53, 95% CI 2-sided [-435.33 to 414.27]
Statistical Analysis 5: Comparison: EDP-305 1 mg vs Placebo; Analysis for C4 AUC0-8; Test type: Superiority; p = 0.412, ANCOVA; Least squares mean difference = -91.7, 95% CI 2-sided [-475.92 to 292.51]
Statistical Analysis 6: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for C4 AUC0-8; Test type: Superiority; p = 0.094, ANCOVA; Least squares mean difference = -250.18, 95% CI 2-sided [-605.33 to 104.98]
Statistical Analysis 7: Comparison: EDP-305 1 mg vs Placebo; Analysis for C4 AUC2-8; Test type: Superiority; p = 0.266, ANCOVA; Least squares mean difference = -83.7, 95% CI 2-sided [-279.15 to 111.75]
Statistical Analysis 8: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for C4 AUC2-8; Test type: Superiority; p = 0.047, ANCOVA; Least squares mean difference = -238.19, 95% CI 2-sided [-470.22 to -6.15]
Statistical Analysis 9: Comparison: EDP-305 1 mg vs Placebo; Analysis for BA AUC0-8; Test type: Superiority; p = 0.694, ANCOVA; Least squares mean difference = 28.41, 95% CI 2-sided [-180.2 to 237.02]
Statistical Analysis 10: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for BA AUC0-8; Test type: Superiority; p = 0.615, ANCOVA; Least squares mean difference = -39.5, 95% CI 2-sided [-264.32 to 185.32]
Statistical Analysis 11: Comparison: EDP-305 1 mg vs Placebo; Analysis for BA AUC2-8; Test type: Superiority; p = 0.974, ANCOVA; Least squares mean difference = 2.93, 95% CI 2-sided [-229.6 to 235.46]
Statistical Analysis 12: Comparison: EDP-305 2.5 mg vs Placebo; Analysis for BA AUC2-8; Test type: Superiority; p = 0.793, ANCOVA; Least squares mean difference = -26.05, 95% CI 2-sided [-283.24 to 231.15]

ADVERSE EVENTS:
Time Frame: Up to 16 Weeks
Arm/Group | EDP-305 1 mg | EDP-305 2.5 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/28 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/31 | 2/28 | 0/9
Other Adverse Events (participants affected / at risk) | 23/31 | 24/28 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-305 1 mg (N=31) | EDP-305 2.5 mg (N=28) | Placebo (N=9)
Headache (Nervous system disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Pruritis (Gastrointestinal disorders) | 0 | 1 | 0
Urticaria (Gastrointestinal disorders) | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | EDP-305 1 mg (N=31) | EDP-305 2.5 mg (N=28) | Placebo (N=9)
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 5 | 3
Paraesthesia (Nervous system disorders) | 1 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 1 | 1
Influenza like illness (General disorders) | 0 | 2 | 0
Swelling (General disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 16 | 3
Pruritus generalised (Skin and subcutaneous tissue disorders) | 5 | 9 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT03394924/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT03394924/SAP_001.pdf